CLINICAL TRIAL: NCT07386028
Title: Full Sternotomy Versus J-shaped Mini-sternotomy for Chronic Ascending Aortic Pathology
Brief Title: Full Sternotomy vs Mini-sternotomy for Ascending Aortic Pathology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk Cardiology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260
Record Dates: First submitted 2025-12-10; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ascending Aortic Aneurysm
Keywords: ascending aortic aneurysm; aortic replacement; sternotomy; mini-sternotomy
MeSH Terms: conditions — Aneurysm, Ascending Aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Sternotomy (Active Comparator): 100 patients who will undergo hemiarch repair via full sternotomy
  Interventions: Procedure: Full sternotomy
- Mini J-Sternotomy (Active Comparator): 100 patients who will undergo hemiarch repair via J-shaped mini-sternotomy
  Interventions: Procedure: J-shaped mini-sternotomy

INTERVENTIONS:
Procedure: Full sternotomy — hemiarch repair via full sternotomy
  Arms: Full Sternotomy
Procedure: J-shaped mini-sternotomy — hemiarch repair via J-shaped mini-sternotomy
  Arms: Mini J-Sternotomy

SUMMARY:
This study investigates outcomes after hemiarch repair in patients with chronic ascending aortic disease. The patients will be divided into two groups according to surgical approach: 100 patients will undergo hemiarch repair via full sternotomy (FS group) and 100 patients will receive hemiarch repair via J-shaped mini-sternotomy (MS group). Early and late outcomes will be recorded.

DETAILED DESCRIPTION:
1. Relevance of the study Hemiarch repair is an effective treatment for patients with ascending aortic aneurysm (AAR). All aortic procedures are routinely performed from full mean sternotomy but nowadays this standard could be performed via minimally invasive approach as well. There are some data that mini-J sternotomy is associated with less blood loss and blood products transfusion, improved lung function and eliminates wound complications risks. The aim of this study was to assess the morbidity and mortality after hemiarch repair via full or J-shaped mini-sternotomy.
2. Patients and methods Patients who will undergo hemiarch repair procedure via full sternotomy (FS group) will be compared with patients who will receive hemiarch repair via J-shaped mini-sternotomy (MS group). Baseline characteristics including preoperative clinical status, details on surgery, and postoperative outcomes will be compared between these groups. Follow-up data will be recorded.

Imaging All aortic measurements will be assessed by electrocardiography-gated computed tomographic angiography. Postoperative computed tomography of the aorta will be performed within 2 weeks after surgery. Analysis will be performed using 64-slice scanner Discovery NM-CT 570c (GE Healthcare, Milwaukee, WI, USA) with spatial resolution of the angiographic phase ranging from 0.6 to 1.25 mm. All measurements will be taken always in the plane perpendicular to the manually corrected local aortic centre line. Ascending aortic diameter will be measured at the level of the pulmonary artery bifurcation. The maximum aortic diameter (mm) will be measured from the outer contours of the aortic wall. All images will be independently assessed by two experienced cardiologists.

Surgical technique The hemiarch repair is performed via a full sternotomy or J-shaped mini-sternotomy under mild-to-moderate hypothermia (28-30°C) and antegrade cerebral perfusion through the innominate artery with side graft. The distal aortic anastomosis is performed using an open anastomosis fashion and involved resection of the inferior portion of the aortic arch from the base of the innominate artery to the projection of the origin of the left subclavian artery. Near infrared spectroscopy (Invos 5100, Somanetics Corp., USA) is used for cerebral monitoring during the operation. When the target temperature is achieved, lower body circulatory arrest with antegrade cerebral perfusion is initiated. The distal aortic anastomosis is performed with a running 4/0 polypropylene suture with a Dacron graft. Proximal aortic reconstruction including Bentall procedure, David procedure, proximal aortic anastomosis, etc. are performed during the rewarming period. The patient is weaned from cardiopulmonary bypass when the body temperature reached 36°C. The sequence of the surgical steps during the operation are the same for all patients.

Follow-up Follow-up will be performed according to the institutional database supplemented by individual patient records. Data will be obtained via medical records of clinical encounters or phone calls with patients and/or relatives. Postoperative computed tomographic scans will be performed upon discharge, at 12 months from the last procedure and at 60 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Ascending aorta greater than 5 cm without involving the aortic arch

Exclusion Criteria:

* Acute aortic dissection or urgent/emergent cases.
* Redo aortic surgery.
* Aortic arch surgery.
* Concomitant CABG or left ventricle restoration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Early mortality | during follow-up time - 60 months
  The difference in the incidence of early mortality between groups (p-value).

SECONDARY OUTCOMES:
Delirium (percent) | Perioperative/Periprocedural
  The difference in the incidence of delirium during follow-up (p-value).
Transient ischemic attack (percent) | Perioperative/Periprocedural
  The difference in the incidence of transient ischemic attack during follow-up (p-value).
Stroke (percent) | during follow-up time - 60 months
  The difference in the incidence of stroke during follow-up (p-value).
Respiratory failure (percent) | Perioperative/Periprocedural
  The difference in the incidence of respiratory failure during follow-up (p-value).
New arrythmia (percent) | during follow-up time - 60 months
  The difference in the incidence of new arrythmia during follow-up (p-value).
Pericardial effusion (percent) | Perioperative/Periprocedural
  The difference in the incidence of new arrythmia during follow-up (p-value).
Heart failure (percent) | during follow-up time - 60 months
  The difference in the incidence of heart failure during follow-up (p-value).
Myocardial infarction (percent) | during follow-up time - 60 months
  The difference in the incidence of myocardial infarction during follow-up (p-value).
Systemic embolism (percent) | during follow-up time - 60 months
  The difference in the incidence of systemic embolism during follow-up (p-value).
Acute kidney injury requiring renal replacement therapy (percent) | during follow-up time - 60 months
  The difference in the incidence of renal replacement therapy during follow-up (p-value).
Re-exploration rate (percent) | during follow-up time - 60 months
  The difference in the incidence of re-operation for bleeding during follow-up (p-value).

CONTACTS AND LOCATIONS:
Overall Officials: Boris N. Kozlov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No